CLINICAL TRIAL: NCT06095700
Title: First Rib Resection Versus Avulsion for the Management of Thoracic Outlet Syndrome
Brief Title: First Rib Resection Versus Avulsion for Thoracic Outlet Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Fahmi Hussein Kakamad, Director of Scientific Department at Smart Health Tower, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UniSulaimani
Record Dates: First submitted 2023-09-15; First posted 2023-10-23 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rib Resection Group (Active Comparator): This arm undergoes first rib resection, as mentioned in the textbook.
  Interventions: Procedure: first rib resection
- Rib Avulsion Group (Experimental): This group of patients undergo first rib avulsion
  Interventions: Procedure: First rib avulsion

INTERVENTIONS:
Procedure: first rib resection — standard first rib resection
  Other Names: surgery
  Arms: Rib Resection Group
Procedure: First rib avulsion — As the active treatment, just instead of resectioning the first rib, we will do an avulsion of the first rib through the same incision
  Arms: Rib Avulsion Group

SUMMARY:
The management of thoracic outlet syndrome can be either surgical or nonsurgical. Fewer than 20% of patients experience benefits from nonsurgical treatments. Regarding the surgical approach, there's considerable debate about whether to resect the first rib or if a scalenectomy alone suffices. Recently, many experts have concurred on the resection of the first rib. Based on our observations, avulsion of the first rib results in improved outcomes and reduced post-operative pain compared to simple resection. Thus, this study aims to compare the outcomes of first rib resection versus its avulsion in patients with thoracic outlet syndrome.

ELIGIBILITY:
Inclusion Criteria: any patient diagnosed as a case of neurogenic thoracic outlet syndrome -

Exclusion Criteria: patients with other types of thoracic outlet syndrome (vascular TOS)

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | six months
  Numeric Rating Scale (NRS) is used to measure satisfaction, the patients are asked to rate their satisfaction on a scale from 0 to 10, with 0 representing "completely dissatisfied" and 10 representing "completely satisfied."
post operative pain | four weeks after the operation
  we use the Visual Analogue Scale. A range of scores from 0-100. A higher score indicates greater pain intensity. the least value is zero and the highest value is 100

CONTACTS AND LOCATIONS:
Overall Officials: fahmi Kakamad, PhD, Study Chair — University of Sulaimani
Locations (1):
- Smart Health Tower, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: Yes